CLINICAL TRIAL: NCT03016780
Title: Evaluation of The Effect of Fecal Microbiota Transplantation on Ulcerative Colitis and Its Mechanism
Brief Title: Fecal Microbiota Transplantation for Ulcerative Colitis
Acronym: FMTFUC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Chengdu Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMT-IBD
Record Dates: First submitted 2017-01-03; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-12

CONDITIONS: Ulcerative Colitis; Intestinal Bacteria Flora Disturbance; Fecal Microbiota Transplantation
Keywords: Ulcerative Colitis; Intestinal Bacteria Flora Disturbance; Fecal Microbiota Transplantation; Intestinal Mucosal Immunity
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment in part 1 (Active Comparator): Fecal microbiota transplantation and traditional treatments will be used in patients with ulcerative colitis in part 1.
  Interventions: Other: Fecal Microbiota Transplantation
- Placebo in part 2 (Placebo Comparator): The traditional treatments and normal saline will be used in patients with ulcerative colitis in part 2 according to associated guidelines.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Other: Fecal Microbiota Transplantation — Fecal microbiota transplantation and the traditional treatments for ulcerative colitis in part 1.
  Other Names: Fecal Microbiota Transplantation(FMT)
  Arms: Treatment in part 1
Other: Normal Saline — Normal saline and the traditional treatments for ulcerative colitisin in part 2.
  Other Names: Normal Saline(NS)
  Arms: Placebo in part 2

SUMMARY:
Ulcerative colitis is a common digestive system disease, the incidence is increasing in recent years.It is reported that the occurrence and development of ulcerative colitis is closely related to imbalance of intestinal flora .Moreover,intestinal mucosal immunity may be related to intestinal flora. Fecal microbiota transplantation as a new technology to rebuild intestinal flora has been used for several disease，but the efficacy of ulcerative colitis by fecal microbiota transplantation needs to be further explored.

DETAILED DESCRIPTION:
Patients who meet the inclusion crit ulcerative colitisby will be separated into two parts depending on accepation or refuse of Fecal microbiota transplantation.Blood specimen from patients will be collected to analysis intestinal mucosal immunity.

ELIGIBILITY:
Inclusion Criteria:

1. subjects voluntarily participate in the trial and sign informed consent;
2. sex is not limited,ranging from 18 to 75 years old;
3. meet the diagnostic criteria for ulcerative colitis in patients;
4. be able to communicate well with the researchers and follow the verification requirements.

Exclusion criteria:

1. Pregnancy or people who are not to give informed consent;
2. use of major immunosuppressive agents, including the use of large doses of glucocorticoids, calcineurin inhibitors, mTOR inhibitors, depleted lymphocyte biological agents, anti-tumor necrosis factor and other conditions; chemotherapy of antineoplastic drugs;
3. decompensated cirrhosis, progressive AIDS and HIV infectionor other serious immunodeficiency disease;
4. use of antibiotics and probiotics within six weeks;
5. with severe complications such as local stenosis, intestinal obstruction, intestinal perforation, toxic colon expansion, colon cancer, rectal cancer patients;
6. combined with cardiovascular, cerebrovascular, liver, kidney and hematopoietic system and other serious primary disease, mental illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 3 months
  According to the inclusion criteria, the patients were randomly divided into experimental group and control group. Before and after the fecal microbiota transplantation, patients were asked about the history of abdominal pain, abdominal distension, diarrhea and so on,at the same time, monitoring heart rate, respiration, pulse, blood pressure is necessary and determinating liver function, renal function, electrolytes, blood coagulation, blood lipids, endotoxins and other biochemical tests to evaluate clinical efficacy.

SECONDARY OUTCOMES:
Improvement of clinical symptoms of the treatment | 4 week
  We evaluate the improvement of clinical symptoms of the treatment through Clinical Symptom Score of ulcerative colitis and Endoscopic Rachmilewitz Scoreto.
The influence of interleukin-10 after the treatment | 0-4 week
  Inflammatory factors such as interleukin-10 in the blood of patients with ulcerative colitis and indicators of disease activity such as erythrocyte sedimentation rate, C-reactive protein are often elevated, we want to study the change above indicators before and after treatment, reflecting the improvement of Inflammation of ulcerative colitis and study the effect of its activity.
Intestinal mucosal immunity | 4 week
  Ulcerative colitis is an autoimmune disease, it is closely related to the secretory SIgA, and content of serum secretory SIgA of ulcerative colitis patients often decreased. By measuring serum secreted SIgA before and after the treatment of to reflect the immune function of ulcerative colitis.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoan Li, Ph.D, Study Chair — First Affiliated Hospital of Chengdu Medical College
Locations (1):
- IEC of Chengdu Medical College, Chendu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tian Y, Zhou Y, Huang S, Li J, Zhao K, Li X, Wen X, Li XA. Fecal microbiota transplantation for ulcerative colitis: a prospective clinical study. BMC Gastroenterol. 2019 Jul 4;19(1):116. doi: 10.1186/s12876-019-1010-4. PMID 31272391